CLINICAL TRIAL: NCT05476172
Title: The Effect of Dienogest vs. Norethindrone Acetate Treatment in Endometriosis
Acronym: DINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8/23
Record Dates: First submitted 2022-07-07; First posted 2022-07-27 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Endometriosis
Keywords: endometriosis; norethindrone acetate; dienogest; chronic pelvic pain; progesterone
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dienogest (Active Comparator): Patients with endometriosis are prescribed dienogest for treatment.
  Interventions: Drug: Dienogest Pill
- Norethindrone Acetate (Active Comparator): Patients with endometriosis are prescribed Norethindrone Acetate for treatment.
  Interventions: Drug: Norethindrone Acetate

INTERVENTIONS:
Drug: Dienogest Pill — The effect of dienogest on endometriosis pain symptoms.
  Other Names: Visanne Group
  Arms: Dienogest
Drug: Norethindrone Acetate — The effect of Norethindrone Acetateon endometriosis pain symptoms.
  Other Names: Primolut-N Group
  Arms: Norethindrone Acetate

SUMMARY:
This randomized controlled study aims to investigate the efficiency of medical treatment modalities in endometriosis patients. The study protocol involves two arms. (Dienogest Group and Noretindrone Acetate Group). The patients diagnosed with endometriosis are randomized depending on their protocol ids. The Dienogest group is prescribed 5 mg dienogest per day and neta group is prescribed 5 mg neta per day. The pain scores will be analyzed six months and twelve months after treatment.

DETAILED DESCRIPTION:
The aim of this observational drug study was to evaluate the patients with medical treatment indications who applied to Bursa Uludağ University Medical Faculty Hospital, Department of Obstetrics and Gynecology, Endometriosis and Chronic Pelvic Pain Outpatient Clinic, during the application of 2 different progesterone protocols with proven efficacy, which are currently recommended for routine use, with 6-month periods and three doses. To compare the effects of different progesterone-derived protocols in use and their effects on treatment effectiveness and recurrence by evaluating ultrasonographic parameters, laboratory parameters, and numerical scoring system scores of patients on chronic pain symptoms (dysmenorrhea, dyspareunia, dysgeusia, and chronic pelvic pain) at different visits.

It was designed as a one-time prospective, randomized observational study. Patients who applied to the Endometriosis and Chronic Pelvic Pain Polyclinic and were evaluated by the relevant faculty members and received medical treatment indications will be randomly assigned to one of the two treatment protocols used as single-digit 'norethindrone acetate' and double-digit 'dienogest' according to the last digit of the current hospital protocol numbers in the system. At the time of the first application, the patients will be recorded in the patient files together with their personal and demographic data, the duration of the previous treatments and the reasons for their discontinuation, the operation notes, and centers of their previous surgeries due to endometriosis, if any. Patients will be evaluated with ultrasonographic evaluations and detailed physical examinations, and laboratory tests. In the ultrasonographic evaluation, uterine contours, presence of adenomyosis, detailed evaluation of the adnexal area, if there is the presence of endometrioma, its size, and the evaluation of the Douglas cavity will be made in detail. Physical examination includes vaginal and rectal examination, and tenderness and nodular appearance will be evaluated. Laboratory parameters include complete blood count, biochemical parameters, tumor markers, and anti-mullerian hormone levels, which we routinely check in the endometriosis outpatient clinic. It will be evaluated and recorded at each visit.

Patients will be questioned for existing dyspareunia, dysmenorrhea, dysgeusia, and chronic pelvic pain. Grades will be written by asking the patients to give a score between 1-10 with the numerical scoring system for their existing pain complaints. In addition, accompanying gastrointestinal and genitourinary symptoms will be noted in the patient's file.

Patients will be reassessed at 6 and 12 months while on treatment with progestins given according to protocol numbers. In addition, at each visit, patients will be evaluated for possible side effects of medical treatment and recorded. In terms of side effects, patients will be asked to give points between 1-10 with the numerical scoring system. Any other side effects will be recorded in the patient file. The information of these records will be taken from the file by the responsible worker after each visit and recorded in the study forms. The study supervisor is not authorized to determine or change the patient's treatment protocol.

In statistical analysis, a comparison between the groups will be made with the Kruskal Wallis test as a non-parametric test using the SPSS-22 program. P value <0.05 will be considered statistically significant.

4. STUDY POPULATION File analysis of all patients between the ages of 18-40 who applied to our center with the diagnosis of endometriosis and met the inclusion criteria will be performed.

CRITERIA FOR INCLUSION

* Patients aged between 18 and 40 who applied to our Endometriosis and Chronic Pelvic Pain Outpatient Clinic
* Patients who do not want pregnancy
* Patients with a diagnosis of endometriosis and a medical suppression indication due to pain.

EXCLUSION CRITERIA

* Patients who are contraindicated to use progesterone
* Patients who have developed an allergic reaction to the progesterone preparations used and the active ingredients in it
* Patients with pelvic inflammatory disease accompanying endometriosis
* Patients diagnosed with uterine malformation with previous surgery
* Patients with obstructive genitourinary and gastrointestinal symptoms and indication for surgical treatment

STUDY CENTER Bursa Uludağ University Faculty of Medicine Hospital, Department of Obstetrics and Gynecology Endometriosis and Chronic Pelvic Pain Polyclinic DETERMINATION OF STUDY POPULATION It is planned to recruit patients between the ages of 18-40 who receive medical treatment indications in Bursa Uludağ University Medical Faculty Hospital, Department of Gynecology and Obstetrics Endometriosis and Chronic Pelvic Pain Polyclinic.

DIAGNOSIS AND TREATMENT PROTOCOL The files of patients who applied to Bursa Uludağ University Gynecology and Obstetrics Department Endometriosis and Chronic Pelvic Pain Polyclinic and started medical treatment will be examined.

The progesterone treatment protocols routinely used in the Endometriosis and Chronic Pelvic Pain Outpatient Clinic are as follows;

1. The use of progesterone, which is started on the second day of the menstrual cycle and continued uninterruptedly (norethindrone acetate 5 mg tablet p.o. 1x1 in posology)
2. Progesterone use, which is started on the second day of the menstrual cycle and continued uninterruptedly (dienogest 2 mg tablet p.o. 1x1 in posology). Apart from the routine operation of the clinic, no non-routine procedures will be performed in the study. The study supervisor does not have the authority to be involved in the treatment and change the protocol. It will only observe and analyze data of treatment protocols initiated from the file.

MATERIALS AND METHODS Patients who applied to the Department of Obstetrics and Gynecology Endometriosis and Chronic Pelvic Pain Polyclinic and received medical suppression treatment indications were included in the study.

No changes will be made in the treatment and follow-up protocols of the patients for the purpose of the study. Patients who are started on medical treatment are routinely called for follow-up at 6-month intervals. At the beginning of the treatment, at the 6th and 12th months of the treatment, all patients will be routinely visited. Patients will not be included in the evaluation of additional controls and examinations for the purpose of the study. The current evaluations of the patients in treatment will be recorded. Patients who are on the protocol of 2 different progesterone derivatives recommended by the guidelines and applied in our clinic will be compared among themselves in terms of laboratory parameters, ultrasonographic evaluations, and numerical scoring systems for chronic pain symptoms, and the effects of these values on treatment effectiveness and recurrence outcomes will be evaluated and the records in the patient files will be examined. The research will be carried out by collecting data from patient files, and the study we have done will not cause any change in the current treatment of patients.

DURATION OF STUDY The duration of the study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years aged women diagnosed with endometriosis

Exclusion Criteria:

* malignancy
* need for surgery
* pregnancy desire

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Chronic Pelvic Pain | Change from Baseline Score at 6 months
  Numeric Score before and after treatment
Chronic Pelvic Pain | Change from Baseline Score at 12 months
  Numeric Score before and after treatment

SECONDARY OUTCOMES:
Side Effect Rate | Rate of Side Effect from baseline at 6 months
  Presence of any side effect related to the drug use
Side Effect Rate | Rate of Side Effect from baseline at 12 months
  Presence of any side effect related to the drug use

CONTACTS AND LOCATIONS:
Overall Officials: Kiper Aslan, Assoc. Prof., Principal Investigator — Uludag University; Isil Kasapoglu, Assoc. Prof., Principal Investigator — Uludag University; Gurkan Uncu, Prof., Study Chair — Uludag University
Locations (1):
- Uludag University, Bursa, Nilufer, Turkey (Türkiye)

REFERENCES:
- [Derived] Gurbuz TB, Aslan K, Kasapoglu I, Muzii L, Uncu G. Norethindrone acetate versus dienogest for pain relief in endometriosis related pain: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2025 Jun;310:113940. doi: 10.1016/j.ejogrb.2025.113940. Epub 2025 Mar 29. PMID 40233572